CLINICAL TRIAL: NCT06887322
Title: The Efficacy of Topical Formulation Containing Ciplukan (Physalis Angulata Linn.) on Modified Psoriasis Area and Severity Index, Thickness, and Inflammation of Psoriasis Vulgaris Lesions
Brief Title: The Efficacy of Topical Formulation Containing Ciplukan (Physalis Angulata Linn.) on Psoriasis Vulgaris Lesions
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DV-202503.01; 1549/UN6.3.1/PT.00/2023 (Other Grant/Funding Number: Universitas Padjadjaran)
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis Vulgaris; Inflammation
Keywords: Physalis angulata Linn.; mPASI; ultrasonography
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bethametasone valerat 0,1% (Active Comparator): A minimum amount of 20 psoriasis vulgaris lesion treated with the bethametasone valerate 0,1% cream, applied twice daily for 14 days.
  Interventions: Drug: Bethametasone valerate 0,1% cream
- Ciplukan (Experimental): A minimum amount of 20 psoriasis vulgaris lesion treated with the topical formulation containing 20% ciplukan (Physalis angulata Linn.) extract, applied twice a day for 14 days.
  Interventions: Drug: Ciplukan

INTERVENTIONS:
Drug: Ciplukan — A minimum amount of 20 psoriasis vulgaris lesion treated with the topical formulation containing 20% ciplukan (Physalis angulata Linn.) extract, applied twice a day for 14 days.
  Arms: Ciplukan
Drug: Bethametasone valerate 0,1% cream — A minimum amount of 20 psoriasis vulgaris lesion treated with the bethametasone valerate 0,1% cream, applied twice daily for 14 days.
  Arms: Bethametasone valerat 0,1%

SUMMARY:
Psoriasis vulgaris is a chronic inflammatory skin disease mediated by the immune system, with a complex pathogenesis that requires long-term therapy. Various inflammatory mediators that activate and are produced from the NF-κB signaling pathway play a role in the pathogenesis of psoriasis vulgaris. Topical corticosteroids are the first-line therapy for all severity levels of psoriasis vulgaris, possessing immunosuppressive, anti-inflammatory, and antimitotic effects. However, long-term use can lead to side effects such as atrophy, striae, telangiectasia, hypopigmentation, acneiform eruptions, perioral dermatitis, and hypertrichosis.

DETAILED DESCRIPTION:
Ciplukan (Physalis angulata Linn.) contains seco-steroids and flavonoids, which exhibit anti-inflammatory, antiproliferative, and immunosuppressive effects. These effects suggest that ciplukan (Physalis angulata Linn.) could serve as an adjuvant topical therapy for psoriasis vulgaris. However, studies on the effectiveness of ciplukan (Physalis angulata Linn.) extract in topical formulations for patients with psoriasis vulgaris have not yet been conducted.

Therefore, a study is needed to assess psoriasis vulgaris lesions both subjectively using the modified PASI score and objectively using high-frequency ultrasonography and spectral Doppler ultrasonography. This would evaluate the effectiveness of ciplukan (Physalis angulata Linn.) cream as an adjuvant topical therapy for psoriasis vulgaris in reducing inflammation and accelerating clinical improvement of skin lesions in patients with psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60 years
* Diagnosed with psoriasis vulgaris based on medical history, physical examination, and severity assessment using the PASI score

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Patients currently undergoing systemic therapy for psoriasis vulgaris.
* Patients who have not discontinued systemic therapy/phototherapy for psoriasis vulgaris ≤ 30 days.
* Patients with psoriasis vulgaris who have not discontinued topical therapy (other than moisturizers) ≤ 14 days.
* Psoriasis vulgaris lesions located in trauma-prone areas, palms, soles, face, and skin folds.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Modified Psoriasis Area and Severity Index (MPASI) | 14 days
  The scoring method that will be used to assess the clinical severity of each observed lesion. The minimum value is 0, and maximum value is 12. A higher scores indicate a worse outcome.
Lesion thickness | 14 days
  High frequency ultrasonography will be used to measure the thickness of each observed lesion (measured in milimeter)
Inflammation | 14 days
  Resistive index detected by high frequency ultrasonography will be used to assess the severity of inflammation in each observed lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Oki Suwarsa, dr., Sp.D.V.E., Subsp.D.A.I., M.Kes, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung; Miranti Pangastuti, dr., Sp.D.V.E., Subsp.D.A.I, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung; Dr. Harry Galuh Nugraha, dr., Sp.Rad(K), Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia